CLINICAL TRIAL: NCT06978660
Title: Multicenter Study for the Validation of an AI-based ECG Platform for Early Cardiac Amyloidosis Diagnosis (CONCERTO)
Brief Title: Multicenter Study for the Validation of an AI-based ECG Platform for Early Cardiac Amyloidosis Diagnosis
Acronym: CONCERTO
Status: Recruiting | Type: Observational
Sponsor: Idoven 1903 S.L. (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: CON_1b
Record Dates: First submitted 2025-05-09; First posted 2025-05-18 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Transthyretin Cardiac Amyloidosis
Keywords: Transthyretin cardiac amyloidosis; ATTR; AI-based ECG Analysis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ATTR-CA patients: Adult patients with confirmed diagnosis of ATTR-CA
- Controls (non ATTR-CA subjects): Adult subjects suspected of ATTR-CA, but finally confirmed not to have ATTR-CA

SUMMARY:
CONCERTO is a retrospective, observational, multicentric and single-arm study to perform an external validation of the cloud-based and AI-powered electrocardiogram (ECG) analysis platform, named Willem™, to detect Transthyretin cardiac amyloidosis (ATTR-CA). Thus, this study will assess Willem™ ability to distinguish between truly diagnosed ATTR-CA patients and confirmed non-ATTR-CA patients from ECG data.

DETAILED DESCRIPTION:
Transthyretin cardiac amyloidosis (ATTR-CA) is an infiltrative cardiomyopathy affecting cardiac health. Results from clinical trials have shown the importance of early diagnosis to improve outcomes and maximize treatment efficacy.

An electrocardiogram (ECG) is the most commonly performed cardiac diagnostic procedure, providing a large amount of information that can reflect cardiac structure and physiology. In this regard, ECG could be an ideal screening tool for ATTR-CA given its wide use, non-invasive nature, low cost and high sensitivity to reflect ATTR-CA abnormalities.

The CE-marked Willem™ ECG Analysis platform has already shown its capability to process ECG data to detect cardiac patterns and arrythmias. This retrospective, observational, multicentric and single-arm study aims to expand the capabilities of the Willem™ ECG Analysis platform, in this case to detect ATTR-CA from ECG analysis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects ≥ 18 years old
* Subjects with 12-leads ECG records with a 10 seconds minimum length on digital format

Exclusion Criteria:

* Patients with paced rhythm on the ECG.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with a suspected or confirmed diagnosis of ATTR-CA
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-05-27 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Device performance | Baseline (closest clinical assessment to ATTR-CA diagnosis)
  Assessment of Willem ability to distinguish between confirmed diagnosed ATTR-CA patients and subjects with no ATTR-CA diagnosis from ECG data of sufficient quality.
  The diagnostic performance metrics will be accuracy, sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV), and F1-score.

SECONDARY OUTCOMES:
Device performance with sub-optimal ECG data quality | Baseline (closest clinical assessment to ATTR-CA diagnosis)
  Assessment of Willem ability to distinguish between confirmed diagnosed ATTR-CA patients and subjects with no ATTR-CA diagnosis from ECG data which does not meet the minimum pre-specified quality requirements.
  The diagnostic performance metrics will be accuracy, sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV), and F1-score.

CONTACTS AND LOCATIONS:
Overall Officials: Pablo García Pavía, MD, PhD, Principal Investigator — Hospital Universitario Puerta de Hierro
Locations (7):
- Northwestern University, Evanston, Illinois, United States
- Centre Hospitalier Universitaire de Toulouse, Toulouse, France
- Italy (2):
  - Careggi University Hospital, Florence
  - United Hospitals of Trieste University Hospital, Trieste
- Spain (3):
  - Hospital Juan Ramón Jiménez, Huelva, Huelva
  - Hospital Universitario Son Llatzer, Palma de Mallorca
  - Hospital Universitario Donostia, San Sebastián

IPD SHARING:
Plan to Share IPD: No